CLINICAL TRIAL: NCT06982482
Title: Artificial Intelligence Based Models for Primary Sjögren's Syndrome Diagnosis Using Laboratory Data: A Chinese Multicenter Retrospective Study
Brief Title: Artificial Intelligence Based Models for Primary Sjögren's Syndrome Diagnosis
Status: Completed | Type: Observational
Sponsor: The Affiliated Nanjing Drum Tower Hospital of Nanjing University Medical School (Other)
Responsible Party: Sponsor
Other Study IDs: B2022-529-04
Record Dates: First submitted 2025-05-13; First posted 2025-05-21 (Actual); Last update posted 2025-05-21 (Actual); Status verified 2025-03

CONDITIONS: Primary Sjögren's Syndrome (pSS)

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
The goal of this observational study is to develop and validate artificial intelligence (AI)-driven models for improving the diagnosis of Primary Sjögren's Syndrome (PSS) using routine laboratory test data. The main question it aims to answer is:

Can AI-based algorithms accurately diagnose Primary Sjögren's Syndrome by analyzing laboratory test results, and do they outperform traditional diagnostic criteria in Chinese populations?

Researchers will retrospectively analyze anonymized clinical records and laboratory data (e.g., autoantibody levels, inflammatory markers) from patients with suspected or confirmed PSS across multiple medical centers in China. No new interventions will be administered, as the study utilizes existing historical data to train and validate the AI models. The performance of AI algorithms will be compared with current diagnostic standards (e.g., ACR/EULAR criteria) in terms of sensitivity, specificity, and clinical utility.

ELIGIBILITY:
Inclusion Criteria:

* Patients with clinician-diagnosed primary Sjögren's syndrome (pSS) meeting the 2016 ACR/EULAR or 2002 ACEG classification criteria (objective oral/ocular dryness, positive anti-SSA/Ro antibodies, or focal lymphocytic sialadenitis on biopsy).
* Control groups: Individuals with non-pSS autoimmune diseases (e.g., rheumatoid arthritis, systemic lupus erythematosus) or non-autoimmune conditions (e.g., dry eye/sicca symptoms without systemic autoimmunity).

Exclusion Criteria:

* Pregnancy, breastfeeding, with a clear diagnosis of other autoimmune diseases, severe infection and malignant tumors.
* Not newly diagnosed in any of the hospitals.
* Without any available laboratory tests.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: This study includes patients with primary Sjögren's syndrome (pSS; diagnosed via 2016 ACR/EULAR or 2002 ACEG criteria: oral/ocular dryness, anti-SSA/Ro+, or positive biopsy) and controls (non-pSS autoimmune diseases or non-autoimmune sicca symptoms). Eligible participants were newly diagnosed at participating hospitals with complete lab data. Exclusions: pregnancy/breastfeeding, other autoimmune diseases, malignancies, severe infections, or missing lab records. Retrospective data spans multicenter clinical records, ensuring real-world validity.
Sampling Method: Probability Sample
Enrollment: 27432 (Actual)
Dates: Start 2013-01-01 (Actual); Primary Completion 2023-01-01 (Actual); Study Completion 2025-01-01 (Actual)

PRIMARY OUTCOMES:
Diagnostic Accuracy of AI Models for Primary Sjögren's Syndrome (pSS) | Data Collection Period: January 1, 2013, to January 31, 2023 (retrospective analysis of historical records). Model Development and Validation: Completed within 12 months of data aggregation.
  The primary outcome measure is the comparative diagnostic accuracy of the AI-driven model versus the 2016 ACR/EULAR classification criteria for PSS. Accuracy will be quantified using sensitivity (true positive rate), specificity (true negative rate), and area under the receiver operating characteristic curve (AUC-ROC). The AI model's performance will be validated against a gold-standard clinician diagnosis based on comprehensive clinical, serological, and histological assessments.

CONTACTS AND LOCATIONS:
Overall Officials: Xinran Yuan, MD, Study Chair — Nanjing Drum Tower Hospital, Affiliated Hospital of Medical School, Nanjing University
Locations (1):
- Nanjing Drum Tower Hospital, Affiliated Hospital of Medical School, Nanjing University, Nanjing, Jiangsu, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Liu S, Wu G, Pan M, Sun Q, Gao C, Long X, Tang C, Yuan X, Sun L. A multi-criterion feature integration framework for accurate diagnosis of Sjogren's disease using routine laboratory tests. NPJ Digit Med. 2025 Nov 27;8(1):729. doi: 10.1038/s41746-025-02110-2. PMID 41310216